CLINICAL TRIAL: NCT02425969
Title: A Randomised Controlled Trial in Stable Intermediate Coronary Lesions and Grey-zone FFR Values With Evaluation of the Diagnostic Utility of Invasive Coronary Physiological Indices and Quantitative Perfusion MRI. The GzFFR Study
Brief Title: A Trial in Stable Intermediate Coronary Lesions and Grey-zone FFR Values
Acronym: GzFFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Golden Jubilee National Hospital (Other Government)
Collaborators: British Heart Foundation (Other); University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GzFFR Protocol Version 2.1
Record Dates: First submitted 2015-03-30; First posted 2015-04-24 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2015-03

CONDITIONS: Grey-zone Fractional Flow Reserve; Intermediate Coronary Lesions; Stable Angina; Coronary Physiology
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimal Medical Therapy (Experimental): Patients will receive secondary prevention and optimal medical therapy to control their anginal symptoms according to international guidelines without PCI of their grey-zone FFR lesion
  Interventions: Drug: Optimal Medical Therapy
- PCI with Optimal Medical Therapy (Active Comparator): Patients will undergo PCI of their grey-zone FFR lesion as well as appropriate secondary prevention. Anti-anginal therapy will be administered as per clinical requirements according to international guidelines.
  Interventions: Procedure: PCI; Drug: Optimal Medical Therapy

INTERVENTIONS:
Procedure: PCI — Patients will have balloon angioplasty and coronary stent insertion for their grey-zone FFR lesion.
  Arms: PCI with Optimal Medical Therapy
Drug: Optimal Medical Therapy — Optimal Medical therapy consists of secondary prevention which will include high dose statin and aspirin as well as anti-anginal therapy according to ESC 2013 international treatment guidelines for stable angina as follows; B-Blocker or Calcium channel blocker as first line agents and Nicorandil or Nitrates or Ranolazine as second line treatment titrated against symptoms to maximum tolerated dose. ACE inhibitors or Angiotensin Receptor Blockers will be prescribed if patients also have a diagnosis of hypertension, LVEF ≤40%, diabetes or CKD where appropriate.

SUMMARY:
In this randomised controlled trial of patients with stable angina and documented intermediate coronary disease with indeterminate or "grey-zone" Fractional Flow Reserve (FFR) we will randomise patients to either optimal medical therapy alone versus optimal medical therapy with PCI and they will be followed up for the primary endpoint of anginal control as measured by the Seattle Angina Questionnaire at 3 months.

DETAILED DESCRIPTION:
Pressure derived fractional flow reserve (FFR) is recognised as being the gold standard method of assessing the physiological significance of angiographically intermediate lesions. A grey-zone exists between the originally validated cut-off for ischemia of <0.75 and the conventionally adopted cut- off of ≤0.80. Pilot data from our centre has suggested that only 1 in 3 coronary arteries with grey-zone FFR values demonstrate myocardial perfusion defects on stress cardiac MRI and others have suggested that the clinical outcomes in patients with grey-zone FFR are favorable with medical therapy alone. As such, stenting all lesions with grey-zone FFR (as currently recommended) may represent over-treatment and could attenuate the overall benefit of an FFR strategy. In addition to this there are flow derived resistance indices of stenosis severity that have superior diagnostic accuracy and may be helpful in correctly classifying patients with grey-zone FFR. In this study we will a comprehensive analysis of lesions with grey-zone FFR values (0.75-0.82 inclusive) using invasive hyperemic pressure, flow and resistance derived indices of severity with quantitative and qualitative 3T perfusion MRI to enable identification of the best invasive predictors of true perfusion defects on 3T cardiac MRI. Patients will be randomised to optimal medical therapy alone versus optimal medical therapy with PCI and followed up for the primary endpoint of anginal control as measured by the Seattle Angina Questionnaire at 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >18 years
2. 30-80% Diameter Stenosis on QCA
3. Stable angina
4. Non ST-elevation myocardial infarction (NSTEMI) with stable symptoms
5. Able to provide informed consent

Exclusion Criteria:

1. STEMI within 5 days
2. Tortuous vessels which would render pressure wire studies difficult or impossible
3. Heavily calcified vessels which would render pressure wire studies difficult or impossible
4. Unstable symptoms requiring definitive interventional management
5. Severe claustrophobia
6. Age >90 years
7. Life expectancy <1 year
8. Estimated Glomerular Filtration Rate <30 mls/min/1.73m2
9. Inability to undergo MRI scanning due to metallic implant or incompatible permanent pacemaker
10. Severe asthma or inability to safely receive an adenosine infusion
11. Left mainstem disease ≤50% or if considered clinically significant by the operating cardiologist either on angiography or intravascular ultrasound.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-04; Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Angina status as per Seattle Angina Questionnaire | 3 months
  Anginal severity as measured by the Seattle Angina Score at 3 months compared with baseline in patients randomized to PCI versus medical therapy.

SECONDARY OUTCOMES:
MACE | 3 and 12 months
  MACE (Death, myocardial infarction, urgent revascularisation and stroke) in patients randomized to PCI versus medical therapy.
Myocardial infarction | 3 and 12 months
  Myocardial infarction in patients randomized to PCI versus medical therapy.
Urgent Revascularisation | 3 and 12 months
  Urgent Revascularisation of the grey-zone FFR lesion in patients randomized to PCI versus medical therapy.
Total number of anti-anginal medications | 3 and 12 months
  Total number of anti-anginal medications in patients randomized to PCI versus medical therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Keith G Oldroyd, M.D., Principal Investigator — National Health Service
Locations (1):
- Golden Jubilee National Hospital, Glasgow, Dunbartonshire, United Kingdom

REFERENCES:
- [Derived] Hennigan B, Berry C, Collison D, Corcoran D, Eteiba H, Good R, McEntegart M, Watkins S, McClure JD, Mangion K, Ford TJ, Petrie MC, Hood S, Rocchiccioli P, Shaukat A, Lindsay M, Oldroyd KG. Percutaneous coronary intervention versus medical therapy in patients with angina and grey-zone fractional flow reserve values: a randomised clinical trial. Heart. 2020 May;106(10):758-764. doi: 10.1136/heartjnl-2019-316075. Epub 2020 Feb 29. PMID 32114516